CLINICAL TRIAL: NCT03961165
Title: BUSCLAB - A Double Blind Randomized Placebo-Controlled Trial Investigating the Effect of Intravenous Butylscopolamine Bromide to Prevent Slow Progress in Labor
Brief Title: BUSCLAB - Buscopan to Prevent Slow Progress in Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Melbye Michelsen, Attending Physician, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/2380
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Labor (Obstetrics)--Complications; Labor; Prolonged, First Stage
MeSH Terms: interventions — Butylscopolammonium Bromide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): 1mL 20 mg/mL butylscopolamine bromide i.v.
  Interventions: Drug: Butylscopolamine Bromide 20 MG/ML
- Placebo (Placebo Comparator): 1mL 9mg/mL NaCl
  Interventions: Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Butylscopolamine Bromide 20 MG/ML — 1 mL Butylscopolamine Bromide 20 mg/mL i.v. Single dose.
  Arms: Treatment arm
Drug: Sodium Chloride 9mg/mL — 1 mL Sodium Chloride 9 mg/mL i.v. Single dose.
  Arms: Placebo

SUMMARY:
To study the effect of Butylscopolamine Bromide on duration of the active phase of first stage of labor in first time mothers who cross the alert-line for labor dystocia, according to the WHO partograph.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Primiparous women
* Spontaneous onset of labor
* Active phase of labor
* ≥37 weeks of gestation
* Vertex position
* Crossing the alert line, i.e. cervical dilatation of less than one cm per hour in the active phase of first stage of labour (cervix dilation ≥3 - <10 cm)
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP and national and local regulations

Exclusion Criteria:

* Multiple gestation
* Elective cesarean section
* Women in labor already receiving oxytocin when crossing the alert line
* Fully dilated cervix when crossing the alert line
* Preeclampsia defined as blood pressure ≥140/90 and proteinuria (1 or more on a urine dipstick on more than one occasion) with debut after 20 weeks of pregnancy
* Known intestinal stenosis, ileus or megacolon
* Persisting maternal tachycardia (heart rate >130 beats per minute)
* Known maternal myasthenia gravis
* Persisting fetal tachycardia (fetal heart rate baseline >170 beats per minute)
* Hypersensitivity to any of the ingredients in IMP or placebo (butylscopolamine bromide or sodium chloride)
* Women with heart disease who are under surveillance with heart rate monitoring during labor
* Known fetal heart disease
* Untreated glaucoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Duration of labor from the time when the participant was given IMP to delivery | Up to 24 hours
  Time to event variable

SECONDARY OUTCOMES:
Duration from when the participant was given IMP, to 10 cm dilatation | Up to 24 hours
  Time to event variable
Mean cervical dilatation rate, calculated as mean cervical dilatation from IMP is given to 10 cm | Up to 24 hours
  Continuous variable
Duration of labor from the onset of active labor (at least 3 cm dilatation) to delivery | Up to 24 hours
  Time to event variable
Spontaneous vaginal delivery vs operative delivery (vacuum, forceps or cesarean delivery) | At birth
  Categorical variable, fraction of all deliveries
Vaginal delivery vs cesarean delivery | At birth
  Categorical variable, fraction of all deliveries
Spontaneous vaginal delivery, vacuum delivery, forceps delivery, or emergency cesarean delivery | At birth
  Categorical variable, fraction of all deliveries
Amount of oxytocin given, measured 1. As total time with treatment | Up to 24 hours
  Continuous variable, minutes
Amount of oxytocin given, measured 2. As International Units (IU) | At birth
  Continuous variable
Pain scores using a Visual Analogue Scale at baseline and 30 minutes after administration of IMP | up to 30 minutes
  Continuous variable, scale 1 to 9, where 9 is most severe pain
Postpartum hemorrhage (mL) | 2 hours after birth
  Continuous variable
Urinary retention, defined as need for urinary catheter before the participants leave the delivery ward | 24 hours after birth
  Categorical variable, fraction of women with urinary retention
Anal sphincter injury | At birth
  Categorical variable, fraction of all deliveries and fraction of all vaginal deliveries
Apgar score at 5 minutes and 10 minutes after delivery | 5 and 10 minutes after birth
  Ordinal variable, score 0 to 10 where 10 is highest score indicating most vital neonate
pH levels in umbilical vein and artery after delivery | At birth
  Continuous variable
Admission to the Neonatal Intensive Care Unit | Within 2 hours after birth
  Categorical variable, fraction of deliveries
Birth experience measured by the validated questionnaire Child Birth Experience Questionnaire | 4 weeks after birth
  Continuous variable for each category

CONTACTS AND LOCATIONS:
Overall Officials: Trond M Michelsen, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaudernack LC, Einarsen AES, Sorbye IK, Lukasse M, Gunnes N, Michelsen TM. The effect of intravenous hyoscine butylbromide on slow progress in labor (BUSCLAB): A double-blind randomized placebo-controlled trial. PLoS Med. 2024 Mar 28;21(3):e1004352. doi: 10.1371/journal.pmed.1004352. eCollection 2024 Mar. PMID 38547322